CLINICAL TRIAL: NCT05186766
Title: The Effect of Video-Assisted Operating Room Introduce Program (VIASP-OR) Developed for Parents on Parental and Child Anxiety: Randomized Controlled Study Protocol
Brief Title: The Effect of Video-Assisted Operating Room Introduce Program (VIASP-OR)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Cafer Özdemir, Head Researcher, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: KAEK-741
Record Dates: First submitted 2021-12-09; First posted 2022-01-11 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Anxiety; Parent-Child Relations
Keywords: Children; Parents; Anxiety; Technology; Video; Surgery
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Video-Assisted Operating Room Introduce Program (VIASP-OR)
  Interventions: Device: Video-Assisted Operating Room Introduce Program
- Control Group (No Intervention): Standart Nursing Care

INTERVENTIONS:
Device: Video-Assisted Operating Room Introduce Program — Video demonstration about operation room
  Other Names: VIASP-OR
  Arms: Intervention Group

SUMMARY:
Aim: The aim of this study is to evaluate the effect of the video-assisted operating room promotion program developed for parents on the anxiety level of parents and children.

Design: Randomized controlled trial. Methods: The participants (N = 80) will be randomly assigned (1:1) to the intervention and control groups using block randomization. In addition to standard care, a video-assisted operating room promotion program, created by fully addressing the perioperative process, will be applied to the participants assigned to the intervention group. Participants in the control group will only receive standard care. Standard care includes verbal information about the surgical process. The sociodemographic and clinical characteristics, along with the anxiety levels of the children and their parents were measured one day before the operation, and the anxiety levels were again measured on the postoperative first and second day.

Discussion: In the literature, it is seen that pediatric surgery personnel can have a beneficial effect in reducing the anxiety of children and their parents. Among these methods, the effectiveness of distraction methods on children's anxiety has also been proven. As for parental anxiety, which can be as important as child anxiety, not enough studies have been done so far, and the existing studies have not been able to come to a decisive conclusion. If parental intervention is found to have positive effects on the child's anxiety in this study are positive, it will contribute to clinical practice and improve clinical outcomes. In this respect, it will fill this gap in the literature.

Impact: This research will add to the evidence for the effectiveness of an intervention that provides parents with visual and auditory information about the process prior to child surgery. It will benefit parents who want to support their children in managing this process. It will also support nurses working in pediatric surgery clinics.

Trial registration: It was registered at ClinicalTrials.gov in December 2021 (…………).

DETAILED DESCRIPTION:
It is a fact that an advanced care process that can provide the necessary support to the parents is needed to reduce the anxiety levels before the surgery. Preparation for surgery for the child and family should focus on their unique needs and include a holistic approach to the child's physical and psychological preparation. For this reason, there is a need for studies that include a holistic approach to managing child and parent anxiety together in line with the family-centered care philosophy. There are different interventions applied to reduce child and parent anxiety in the preoperative process. Examples of these interventions are simply explaining complex information to parents by visualizing data via a tablet computer, clown intervention, distraction through music, humor, therapeutic play, and audio-visual methods. Introducing the real operating room environment, which is full of unknowns and other than traditional education methods, with video can have a positive effect on reducing the anxiety of parents and children. For this reason, we think that such a study will make a positive contribution to the literature.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children aged 7-12
* Parents whose child will undergo surgery for the first time
* Parents of children who will undergo elective surgery
* Parents who can speak Turkish, understand what they read and listen to, and can apply what is said will be included.

Exclusion Criteria:

* Parents with previous surgical experience
* Parents who used psychiatric drugs
* Parents with a child receiving sedative premedication

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Parent Anxiety- | First day before operation
  The State Anxiety Inventory (STAI-S) The scores obtained from this scale range from a minimum of 20 to a maximum of 80. High score means high anxiety level and low score means low anxiety level.
Parent Anxiety | First day after operation
  The State Anxiety Inventory (STAI-S) The scores obtained from this scale range from a minimum of 20 to a maximum of 80. High score means high anxiety level and low score means low anxiety level.
Parent Anxiety | Second day after operation
  The State Anxiety Inventory (STAI-S) The scores obtained from this scale range from a minimum of 20 to a maximum of 80. High score means high anxiety level and low score means low anxiety level.

SECONDARY OUTCOMES:
Child anxiety | First day before operation
  Facial Affective Scale (FAS) The FAS used for children consists of 5 facial expressions. In expressions ranging from 1 to 5, the first facial expression indicates no anxiety, and the fifth facial expression indicates a very high level of anxiety.
Child anxiety | First day after operation
  Facial Affective Scale (FAS) The FAS used for children consists of 5 facial expressions. In expressions ranging from 1 to 5, the first facial expression indicates no anxiety, and the fifth facial expression indicates a very high level of anxiety.
Child anxiety | Second day after operation
  Facial Affective Scale (FAS) The FAS used for children consists of 5 facial expressions. In expressions ranging from 1 to 5, the first facial expression indicates no anxiety, and the fifth facial expression indicates a very high level of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru KARAZEYBEK, Study Director — Akdeniz University Faculty of Nursing; Aysegul ISLER DALGIC, Study Director — Akdeniz University Faculty of Nursing
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ozdemir C, Duzgun MV, Karazeybek E, Isler Dalgic A. The effect of a video-assisted operating room promotion program on the anxiety levels of parents and their children: A randomized controlled trial protocol. J Pediatr Nurs. 2022 Nov-Dec;67:e150-e155. doi: 10.1016/j.pedn.2022.08.006. Epub 2022 Aug 19. PMID 35995689